CLINICAL TRIAL: NCT00178243
Title: A Phase I/II Trial Of the Feasibility of Treatment of Cancer Involving the Liver With High Dose Radiation Delivered by 3D Conformal Radiation Therapy and Radiosurgery
Brief Title: Feasibility of Treatment of Cancer Involving the Liver With High Dose Radiation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URCC 2298
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2006-09

CONDITIONS: Liver Neoplasms; Neoplasm Metastasis
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis | interventions — Radiotherapy, Conformal; Radiosurgery

INTERVENTIONS:
Procedure: 3D Conformal Radiation Therapy and Radiosurgery

SUMMARY:
A study is being conducted by the University of Rochester Cancer Center (URCC) in which patients with liver cancer will be treated with high dose conformal radiation therapy. This type of radiation uses new techniques which aim the radiation to the sites of disease allowing the tumor to receive a high dose and the surrounding normal liver tissue to receive a low enough dose that the normal tissue should remain free from injury.

The purpose of the study is to determine if the conformal radiation therapy is safe, tolerable and effective in treating liver cancer and to determine the side effects caused by this treatment. A second objective is to determine if the levels of a special type of protein (called cytokines) found in the blood are related to this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have new hepatic lesions suggestive of metastasis, or otherwise biopsy proven disease if there is no previously negative scan.
* Patients with chemotherapy responsive or resistant disease are acceptable. Primary hepatobiliary tumors are also acceptable. In each case, the patient must be deemed unresectable by a hepatic surgeon.
* Patients with multiple hepatic lesions may be included if they meet the volumetric criteria for dose specification. Likewise, patients with metastases to organs other than the liver, or patients with residual primary disease may be included if it is judged that longevity will be determined by the hepatic disease.
* KPS ≥70
* Age ≥ 18 years
* Bilirubin <2.0 mg/dl, AST < 2.5 x normal, ALT < 2.5 x normal, Platelets > 80,000/mm3
* Chemotherapy treatment before or after radiation will be allowed
* Informed consent must be obtained., Patient must be judged unresectable by a hepatic surgeon, or must have refused surgery
* Patient must be able to tolerate radiation treatment as judged by the Principal Investigator or co-PI.
* Previous Liver resection is allowed
* Active disease outside the liver is allowed.
* Liver lesion should be visible on CT or MRI.

Exclusion Criteria:

* No active hepatitis or radiographic evidence of diffuse macro-nodular cirrhosis. Patients with lesser degrees of cirrhosis, not associated with portal hypertension or hepatic failure, are eligible but radiation schedule and total dose will be appropriately modified.
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Paul Okunieff, MD, Principal Investigator — Universtiy of Rochester, Dept of Radiation Oncology
Locations (1):
- University of Rochester, Dept. Radiation Oncology, Rochester, New York, United States